CLINICAL TRIAL: NCT05134610
Title: Effectiveness of Perioperative Oscillating Positive Expiratory Pressure (OPEP) Therapy in Reduction of Post-operative Respiratory Morbidity in Patients Undergoing Colorectal Surgery: a Pilot Randomized Control Trial
Brief Title: Effect of Perioperative OPEP Therapy on Post-operative Pulmonary Complications
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Nawar Alkhamesi MD, Principle Investigator, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 116736
Record Dates: First submitted 2021-11-14; First posted 2021-11-26 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Pulmonary Complication; Surgery--Complications; Surgery
Keywords: oscillating pulmonary expiratory pressure therapy; OPEP

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control (No Intervention): Standard of care for pre- and post-op pulmonary care
- OPEP Therapy (Experimental): 14 days pre- and and post-op OPEP device usage
  Interventions: Device: AEROBIKA POSITIVE EXPIRATORY PRESSURE DEVICE

INTERVENTIONS:
Device: AEROBIKA POSITIVE EXPIRATORY PRESSURE DEVICE — Intervention arm patients use the OPEP device twice daily for 2 weeks before and after surgery
  Arms: OPEP Therapy

SUMMARY:
For patients undergoing colorectal surgery, post-operative pulmonary complications (PPCs) are common. PPCs are associated with increased morbidity and mortality, as well as prolonged hospital stays and healthcare costs. Pulmonary exercise in the pre-operative setting is thought to improve pulmonary fitness and decrease incidence of PPCs. Use of an oscillating positive expiratory pressure (OPEP) device sees patients improve their respiratory fitness through prescribed usage of a handheld instrument that exercises pulmonary muscles while breathing. Here, the investigators propose a pilot randomized-controlled trial (RCT) to evaluate the feasibility of a large scale study that would examine the effect of preoperative OPEP device exercises in preventing PPCs for patients undergoing elective colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years of age or older, and scheduled for an elective colorectal procedure at London Health Science Center (LHSC). Informed consent must be obtained.

Exclusion Criteria:

* Patients unable to perform written consent will be excluded. The investigators will not include colorectal procedures performed for urgent or emergent indications. Patients with advanced pulmonary disease necessitating home oxygen pre-operatively will be excluded. Patients that are pregnant will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Trial feasibility: capacity for recruitment | 18 months
  Ability of clinics to recruit patients in a timely manner. To be reported as a percent of the desired number of patients recruited over an 18 month period.
Trial feasibility: device adherence | 18 months
  Adherence of enrolled patients to usage of the OPEP device. To be reported as percent of patients returning a complete logbook detailing their consistent use of the OPEP device pre-op and post-op.
Trial feasibility: data collection | 18 months
  3) Completeness of data collected from enrolled patients medical record. To be reported as a percent of recruited patients with complete datasets following the trials completion. Used to identify gaps in data for a future fully powered trial.
Trial feasibility: limited efficacy of the OPEP device | 18 months
  Limited efficacy of the OPEP device to decrease post-operative pulmonary complications (PPCs). PPCs represents a composite outcome including atelectasis, pneumonia, prolonged requirement for supplemental oxygen, and respiratory failure.

IPD SHARING:
Plan to Share IPD: Undecided